CLINICAL TRIAL: NCT01232829
Title: A Phase II Study of the Gamma Secretase Inhibitor RO4929097 in Previously Treated Metastatic Pancreas Cancer
Brief Title: Gamma Secretase Inhibitor RO4929097 in Previously Treated Metastatic Pancreas Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02537; NCI-2011-02537 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000687335; 10-0273 (Other: Colorado Multiple Institutional Review Board); 8490 (Other: CTEP); U01CA070095 (NIH); P30CA046934 (NIH)
Record Dates: First submitted 2010-10-30; First posted 2010-11-02 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-06

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (RO4929097) (Experimental): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Patients may undergo tumor biopsy at baseline and on days 16 or 17 of course one for biomarker and other correlative studies. Blood samples may also collected at baseline and periodically during study for pharmacokinetic and angiogenesis marker studies.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given PO
  Other Names: R4733; RO4929097

SUMMARY:
This phase II trial is studying how well RO4929097 (gamma-secretase/Notch signalling pathway inhibitor RO4929097) works in treating patients with previously treated metastatic pancreatic cancer. RO4929097 may stop the growth of tumor cells by blocking some enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 6-month survival of patients with previously treated metastatic pancreas cancer treated with gamma secretase RO4929097.

II. To determine the adverse events of RO4929097 in this patient population. III. To correlate changes in tumor markers with RO4929097 exposure.

SECONDARY OBJECTIVES:

I. To evaluate the response rate and overall survival of this population treated with RO4929097.

II. To correlate clinical outcome with tumor markers (including stem cell markers) obtained from pre- and post- treatment biopsies. (exploratory) III. To assess variants in genes involved in RO4929097 disposition and their relation to RO4929097 exposure.

OUTLINE: This is a multicenter study.

Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 orally (PO) once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

Patients may undergo tumor biopsy at baseline and on days 16 or 17 of course one for biomarker and other correlative studies. Blood samples may also collected at baseline and periodically during study for pharmacokinetic and angiogenesis marker studies.

After completion of study therapy, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma

  * Not amenable to potentially curative surgical resection
* At least 1 prior regimen of chemotherapy, preferably gemcitabine-based, for metastatic disease

  * Evidence of disease progression
* Measurable disease defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan
* Available archived tumor tissue (baseline core biopsies or surgical tumor blocks)

  * No diagnosis by fine-needle aspiration only
* No known brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 (Karnofsky 70-100%)
* White blood cell count (WBC) ≥ 3,000/mm³
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin normal
* Aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Willingness to undergo 2 tumor biopsies, if required
* Fertile patients must use 2 forms of contraception (i.e., barrier contraception and one other method of contraception) ≥ 4 weeks prior to, during, and for ≥ 12 months after completion of therapy
* Negative pregnancy test
* Not pregnant or nursing
* Able to swallow pills
* No patients with malabsorption syndrome or other condition that would interfere with intestinal absorption
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma secretase inhibitor RO4929097
* Not serologically positive for hepatitis A, B, or C
* No history of liver disease, other forms of hepatitis, or cirrhosis
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia despite adequate electrolyte supplementation
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia other than chronic, stable atrial fibrillation
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* No other malignancy within the past 5 years except curatively treated basal cell carcinoma of the skin or carcinoma in-situ of the uterine cervix
* No combination antiretroviral therapy for HIV-positive patients
* Recovered to < Common Toxicity Criteria for Adverse Effects (NCI CTCAE) grade 2 toxicities from prior therapy
* More than 3 weeks since prior chemotherapy for metastatic disease (6 weeks for carmustine or mitomycin C)
* At least 4 weeks since prior radiotherapy
* Concurrent low-molecular weight heparin (LMWH) or full-dose coumadin allowed

  * International normalized ratio (INR) must be monitored as clinically indicated
* No other concurrent investigational agents
* No concurrent strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers, including the following:

  * Strong inhibitors: Amiodarone, erythromycin, clarithromycin, grapefruit juice, isoniazid, ketoconazole, itraconazole, or nefazodone

    * Patients taken off strong inhibitors allowed provided they have ≥ 1-week washout period
  * Strong inducers: Carbamazepine, pentobarbital, phenobarbital, phenytoin, Rifabutin, Rifampin, or St. John wort

    * Patients taken off strong inducers allowed provided they have ≥ 2-week washout period
* No concurrent antiarrhythmics or other medications known to prolong QTc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, Principal Investigator — University of Colorado Cancer Center - Anschutz Cancer Pavilion
Locations (3):
- United States (3):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado, Denver, Colorado
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase II, single-arm study. From December 2010 to May 2012, a total of eighteen patients were enrolled at the University of Colorado Cancer Center and Johns Hopkins Hospital.
Pre-assignment Details: Subjects were eligible if they were at least 18 years old, had a Karnofsky Performance Status of ≥70, at least one previous chemotherapy for metastatic disease, histologically or cytologically metastatic adenocarcinoma of the pancreas, and measurable disease. Patients with islet cell neoplasms and locally advanced disease were excluded.
Groups:
- Treatment (RO4929097): RO4929097 was administered at a dose of 20 mg daily on days 1-3, 8-10 and 15-17 of 21-day cycles.
Period: Overall Study
Arm/Group | Treatment (RO4929097)
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A patient that is alive at 6 months is considered a treatment success. The largest success proportion where the proposed treatment was considered ineffective was 15% and the smallest was 35%. This MinMax design used 32 patients to test the null hypothesis that the true success proportion in a given patient population is at most 15%.
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate
Description: The primary endpoint of the study was 6-month survival. The proportion of successes was estimated by the number of successes divided by the total number of evaluable patients.
Time Frame: 6 months
Population: All patients meeting the eligibility criteria and who received treatment were considered evaluable for the primary endpoint. All patients treated per protocol (n=18) were evaluable for the 6-month survival endpoint.
Measure: Number; unit: participants
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 18
participants | 5

2. Secondary Outcome: Survival
Description: Survival was estimated using the Kaplan-Meier (1958) method.
Time Frame: From registration to death due to any cause, assessed up to 2 years
Population: All patients meeting the eligibility criteria and who received treatment per protocol (n=18) were evaluable for the overall survival endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 18
months | 4.1 [2.7 to 5.8]

3. Secondary Outcome: Time to Disease Progression
Description: Eighteen patients were evaluable for the time to disease progression endpoint.
Time Frame: From registration to documentation of disease progression, assessed up to 2 years
Population: All patients meeting the eligibility criteria and who received treatment per protocol (n=18) were evaluable for the progression-free survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 18
months | 1.5 [1.3 to 1.6]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed within 21 days of receiving the study drug.
Description: Within the 21 days of receiving the study drug, routine blood tests and physical examinations were done.
Arm/Group | Treatment (RO4929097)
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (RO4929097) (N=18)
Confusion (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (RO4929097) (N=18)
Hyperglycemia (Metabolism and nutrition disorders) | 2
Fatigue (General disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Lymphocyte Count Decreased (Investigations) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
The study met criteria to accrue 32 subjects but only 18 were enrolled. It was decided to stop further enrollment after RO4929097 was discontinued by the sponsor and was no longer a development candidate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less